CLINICAL TRIAL: NCT04302649
Title: Influence of Dialysate Temperature on Peritoneal Creatinine Clearance in Patients in Peritoneal Dialysis
Brief Title: Dialysate Temperature in Peritoneal Dialysis
Acronym: TPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Gianni Cappelli, Professor, Azienda Ospedaliero-Universitaria di Modena
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 165/2018/SPER/AOUMO
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Peritoneal Dialysis Complication
Keywords: peritoneal dialysis; dialysate temperature; peritoneal creatinine clearance

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group (Experimental): Patients received Peritoneal Equilibration Test (PET). In the intervention group, dialysate was warmed in a specific microwave oven calibrated to 37°C and infusion temperature was confirmed to be 37°C before infusion
  Interventions: Drug: peritoneal dialysate at 37°C temperature
- Control group (No Intervention): Patients received Peritoneal Equilibration Test (PET). In the control group, current practice was used (batch warming with a pad calibrated to 37°C) and dialysate temperature was measured just before infusion.

INTERVENTIONS:
Drug: peritoneal dialysate at 37°C temperature — during a PET test, patients received peritoneal dialysate warmed at 37°C before infusion
  Arms: Intervention group

SUMMARY:
Patients on continuous ambulatory peritoneal dialysis (PD) are encouraged to warm dialysate to 37°C before peritoneal infusion; main international PD guidelines do not provide specific recommendation, and patients generally warm dialysate batches partially or do not warm them at all. Warming of dialysate is a time-consuming procedure, not free from potential risks (i.e. degradation of glucose), and should be justified by a clear clinical benefit. The investigators designed a single blind randomized controlled trial where PD patients were randomized to receive a peritoneal equilibration test either with dialysate at a controlled temperature of 37°C (intervention group) or with dialysate warmed with conventional methods (control group). Primary end-point was a higher peritoneal creatinine clearance in patients in the intervention group.

DETAILED DESCRIPTION:
Peritoneal dialysis (PD) currently represents the main choice for home renal replacement treatment for patients with end stage renal disease. One of the limitations of PD technique is represented by the difficulty in achieving target dialytic clearances and PD adequacy for some patients, especially with increasing PD vintage. A potentially relevant issue in PD clearances is the effect of dialysate temperature on depuration. Indeed, it is common for clinicians to advise patients in Continuous Ambulatory Peritoneal Dialysis (CAPD) to warm the dialysate before infusion into the peritoneal cavity, with different methods (microwave oven, warming cabin, warming pad). Nevertheless, main international PD guidelines do not provide specific recommendations on this topic. Only guidelines from the British Columbia Renal Agency (Canada) dedicate a specific chapter to the temperature of dialysate, recommending its warming to 37°C before peritoneal infusion, mainly in order to avoid an "uncomfortable lowering of body temperature". On the other hand, warming of PD batches could lead to hot spots formation inside the batch, especially with microwaves, and to degradation of glucose leading to the formation of toxic glucose degradation products (GDPs). Also, notable differences in room temperature exist according to geographical latitude and year season, and there are no clear and detailed reports in the literature regarding intolerable effects of the infusion of dialysate at room temperature. It must be acknowledged that it is common practice for patients to warm dialysate batches only partially or not to warm them at all. Moreover, warming pads that are most commonly used by CAPD patients do not effectively warm the dialysate up to 37°C. In the Peritoneal Dialysis Unit at Azienda Ospedaliero-Universitaria di Modena, it was recently observed that average dialysate temperature at infusion was 31.1°C, even if the pad was calibrated to 37°C [unpublished data]. With respect to the effects on toxins clearances through the peritoneal membrane, a higher dialysate temperature could theoretically favor vasodilation of peritoneal membrane microcirculation, potentially increasing the passage of substances. Severe microcirculatory dysfunction has been reported in PD patients and any intervention designed to ameliorate microcirculatory flow at peritoneal level could be beneficial. Surprisingly, reports regarding the effects of dialysate temperature on peritoneal clearances in PD in humans are surprisingly scarce. In 1967 Gross et al reported an increase in the exchange of substances between peritoneal fluid and blood upon warming of the PD fluid to 37°C (compared to 20°C) in a patient treated with intermittent peritoneal dialysis; the increase in urea clearance with the 37°C solution was 35% on average. In contrast, Indraprasit et al did not encounter differences in peritoneal creatinine clearance utilizing dialysate at room temperature (27-31°C) and warmed at 37°C in a group of 18 patients in PD. Confirmation of the effects of dialysate temperature on peritoneal clearances would be of great interest in order to maximize the depurative potential of PD and to justify patients' effort to warm the batches.

In order to determine the real effects of dialysate temperature on peritoneal clearances and transport characteristics, abdominal discomfort and vital signs, the investigators designed a randomized controlled trial comparing two strategies of peritoneal dialysate warming.

Study design and participants PD patients, both in CAPD and automated PD, in regular follow-up at the Nephrology Unit of the University Hospital of Modena, were randomized to receive a single dialysis exchange, either with dialysate at a controlled temperature of 37°C (intervention group) or with dialysate at warmed with conventional methods at uncontrolled temperature (control group). Randomization was generated through the use of the Random Allocation software11.

Primary end-point of our study was peritoneal creatinine clearance. Secondary end-points were: peritoneal urea clearance, creatinine and urea mass transfer area coefficient (MTAC), abdominal discomfort, blood pressure and body temperature.

A power analysis was performed while designing the study using the few data available in the literature; setting the alpha-error level at 0.05 for a 2-tailed t-test with a statistical power of 95% (beta-error 0.05) the estimated sample needed was 14 patients (7 per group).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* ability to give informed consent
* peritoneal dialysis (PD) treatment
* PD vintage of more than 3 months
* absence of signs of active acute systemic or localized infections at least four weeks apart from the trial

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
peritoneal creatinine clearance | 4 hours - Peritoneal equilibration test
  Peritoneal clearance of creatinine was calculated with the following formula:
  Cx = [Dx] x dialysate volume / [Px] / 240 where Cx represents clearance of creatinine expressed in ml/min, [Dx] represents the concentration of creatinine in dialysate at the end of the exchange (4 hours) expressed in mg/dl, dialysate volume represents the total volume drained at the end of the exchange (4 hours), [Px] represents the concentration of creatinine in plasma after 2 hours from the beginning of the exchange expressed in mg/dl and 240 represents minutes contained in the 4 hours of the exchange.

SECONDARY OUTCOMES:
peritoneal urea clearance | 4 hours - Peritoneal equilibration test
  Peritoneal clearance of urea was calculated with the following formula:
  Cx = [Dx] x dialysate volume / [Px] / 240 where Cx represents clearance of urea expressed in ml/min, [Dx] represents the concentration of urea in dialysate at the end of the exchange (4 hours) expressed in mg/dl, dialysate volume represents the total volume drained at the end of the exchange (4 hours), [Px] represents the concentration of urea in plasma after 2 hours from the beginning of the exchange expressed in mg/dl and 240 represents minutes contained in the 4 hours of the exchange.
creatinine and urea mass transfer area coefficient | 4 hours - Peritoneal equilibration test
  Mass transfer area coefficients (MTAC) for creatinine and urea were calculated with the RenalSoft software (converted from the PD Adequest software) from Baxter Healthcare, Deerfield, IL, U.S.A. Correction for plasmatic water concentration was not added, since the main purpose was to compare MTACs from the intervention and control group and not to obtain absolute data.

CONTACTS AND LOCATIONS:
Overall Officials: Gianni Cappelli, Professor, Principal Investigator — University of Modena and Reggio Emilia
Locations (1):
- Azienda Ospedaliera Universitaria di Modena, Modena, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez-Reyes MJ, Bajo MA, Del Peso G, Ossorio M, Diaz R, Carretero B, Selgas R. The influence of initial peritoneal transport characteristics, inflammation, and high glucose exposure on prognosis for peritoneal membrane function. Perit Dial Int. 2012 Nov-Dec;32(6):636-44. doi: 10.3747/pdi.2011.00137. Epub 2012 Apr 2. PMID 22473036
- [Background] Bargman JM, Krediet RT, Lo WK, Selgas R, del Peso G, Auxiliadora Bajo M, Mujais S. What are the problems with using the peritoneal membrane for long-term dialysis? Semin Dial. 2008 Jan-Feb;21(1):11-23. doi: 10.1111/j.1525-139X.2007.00385_1.x. No abstract available. PMID 18251949
- [Background] Aroeira LS, Aguilera A, Sanchez-Tomero JA, Bajo MA, del Peso G, Jimenez-Heffernan JA, Selgas R, Lopez-Cabrera M. Epithelial to mesenchymal transition and peritoneal membrane failure in peritoneal dialysis patients: pathologic significance and potential therapeutic interventions. J Am Soc Nephrol. 2007 Jul;18(7):2004-13. doi: 10.1681/ASN.2006111292. Epub 2007 Jun 13. PMID 17568021
- [Background] Dombros N, Dratwa M, Feriani M, Gokal R, Heimburger O, Krediet R, Plum J, Rodrigues A, Selgas R, Struijk D, Verger C; EBPG Expert Group on Peritoneal Dialysis. European best practice guidelines for peritoneal dialysis. 7 Adequacy of peritoneal dialysis. Nephrol Dial Transplant. 2005 Dec;20 Suppl 9:ix24-ix27. doi: 10.1093/ndt/gfi1121. No abstract available. PMID 16263748
- [Background] Welten AG, Schalkwijk CG, ter Wee PM, Meijer S, van den Born J, Beelen RJ. Single exposure of mesothelial cells to glucose degradation products (GDPs) yields early advanced glycation end-products (AGEs) and a proinflammatory response. Perit Dial Int. 2003 May-Jun;23(3):213-21. PMID 12938820
- [Background] Fontana F, Ballestri M, Makomi C, Morandi R, Cappelli G. Hemorheologic alterations in peritoneal dialysis. Clin Hemorheol Microcirc. 2017;65(2):175-183. doi: 10.3233/CH-16152. PMID 27340762
- [Background] Gross M, McDonald HP Jr. Effect of dialysate temperature and flow rate on peritoneal clearance. JAMA. 1967 Oct 23;202(4):363-5. No abstract available. PMID 6072310
- [Background] Indraprasit S, Namwongprom A, Sooksriwongse C, Buri PS. Effect of dialysate temperature on peritoneal clearances. Nephron. 1983;34(1):45-7. doi: 10.1159/000182977. PMID 6855994
- [Background] Saghaei M. Random allocation software for parallel group randomized trials. BMC Med Res Methodol. 2004 Nov 9;4:26. doi: 10.1186/1471-2288-4-26. PMID 15535880
- [Background] Teixido-Planas J. Peritoneal function and adequacy calculations: current programs versus PD Adequest 2.0. Perit Dial Int. 2002 May-Jun;22(3):386-93. PMID 12227398
- [Background] Figueiredo AE, Goodlad C, Clemenger M, Haddoub SS, McGrory J, Pryde K, Tonkins E, Hisole N, Brown EA. Evaluation of physical symptoms in patients on peritoneal dialysis. Int J Nephrol. 2012;2012:305424. doi: 10.1155/2012/305424. Epub 2012 Sep 25. PMID 23050149
- [Background] Twardowski ZJ. Clinical value of standardized equilibration tests in CAPD patients. Blood Purif. 1989;7(2-3):95-108. doi: 10.1159/000169582. PMID 2663040
- [Derived] Fontana F, Torelli C, Giovanella S, Ligabue G, Alfano G, Gerritsen K, Selgas R, Cappelli G. Influence of dialysate temperature on creatinine peritoneal clearance in peritoneal dialysis patients: a randomized trial. BMC Nephrol. 2020 Oct 27;21(1):448. doi: 10.1186/s12882-020-02113-z. PMID 33109094